CLINICAL TRIAL: NCT04261101
Title: Test-enhanced Learning Using Causal Connections to Prepare for Future Learning in Endocrinology: a Randomized Clinical Trial
Brief Title: Test-enhanced Learning to Prepare for Future Learning in Endocrinology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 26118919.6.0000.5327
Record Dates: First submitted 2020-01-31; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Endocrinopathy; Educational Problems
MeSH Terms: conditions — Endocrine System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block A (Experimental): Test intervention with questions regarding diabetes and adrenal
  Interventions: Other: Test-enhanced learning
- Block B (Active Comparator): Test intervention with questions regarding thyroid and hypophysis
  Interventions: Other: Test-enhanced learning

INTERVENTIONS:
Other: Test-enhanced learning — Test-enhanced learning with short answers of questions regarding diabetes and adrenal

SUMMARY:
The use of test-enhanced learning with causal connection and in preparation for future learning has been used in health educational setting with positive results. However, most studies were performed in a controlled lab scenario and not in the "real world" of medicine classes, decreasing the external applicability of such experiments. Therefore, the aim of present study is to evaluate if a session of test-enhanced learning at the beginning of endocrinology course, using basic-clinical sciences connections of key concepts, would prepare for future learning of endocrinology on a theory-practical 4-week endocrinology course.

Methods Study design, participants and description of undergraduate endocrinology course This is a prospective, single center, non-blinded, RCT. Participants are students of medicine from Universidade Federal do Rio Grande do Sul (UFRGS), Brazil, in their third year of Medical School, recruited at the beginning of endocrinology undergraduate clinical placement. This clinical trial follows the Consolidated Standards of Reporting Trials (CONSORT) statement, which includes the completing the CONSORT checklist.

Sample size Based in a previous study, to find a difference in the percentage of correct answers in a cognitive test to evaluate retention of 12%, considering a SD of 26%, alpha error of 5%, beta error of 20%, and repeated assessments (baseline, 3 weeks and 6 months), 35 students will be necessary in each group. To account for possible losses of follow-up, 84 students will be included.

Study intervention All students will receive, in advance, a text with basic sciences information relevant to the learning of Endocrinology (supplementary material), with instructions to study the text before intervention day.

Students will be randomized to one of the interventions: TEL with questions about diabetes and adrenal (Block A, 6 questions) or thyroid and hypophysis (Block B, 6 questions). Important endocrinology concepts, such as fuel metabolism and circadian rhythm will be included in Block A, and feedback loops and hormone synthesis in Block B. Specific hormone functions will be part of both TEL Blocks.

Assessments At the same day of intervention, students will answer all questions 12 of the TEL session (questions from blocks A and B) with best answer multiple choice questions (immediate retention test). After 3 weeks and 6 months, the transfer of knowledge will be assessed with a 24 multiple choice questions test, based in clinical cases.

DETAILED DESCRIPTION:
Introduction The ability to connect previous learned basic-sciences concepts to patient's clinical features can help improve clinical reasoning. While experts use several shortcuts to reach a correct diagnosis, such as clinical presentation patterns, "stored" due to years of exposure to real cases, the novice need other strategies to build diagnostic scripts to achieve expertise. Inexperienced medical students acquire clinical reasoning by exploring why specific symptoms occur, usually based on basic science mechanisms. Even experienced physicians apply these connections to solve difficult cases, though sometimes, not in a conscious way. Benefits of causal connections between basic and clinical sciences for clinical reasoning is supported by randomized clinical trials (RCTs). When teaching endocrinology, this strategy acquires additional relevance, as basic concepts regarding hormone action and regulation (ex: feedback loops) are commonly utilized in day-to-day patient care.

Test-enhanced learning is an effective strategy to optimize knowledge acquisition, through formative assessment with the sole objective to promote learning. Testing improves learning through two means: a) an indirect benefit, as it stimulates preparation for the test, and b) through a direct effect, in which the mental effort to answer a question mobilizes and brain connections and reinforces learning. This educational tool has been studied in health professions education, including medical school and clinical training. The utilization of test-enhanced learning with short answers is more efficacious than only restudy or self-explanation. Moreover, the effect lasted for at least 6 months.

More important than content retention and linkage between biomedical concepts and clinical features, is the idea that knowledge must be applied in a different context in the future, a capacity named adaptive expertise. An essential part of training for adaptive expertise is preparation for future learning. It means that a learning session should prepare the student for future acquisition of content, competences and abilities. Medicine is certainly an area where adaptive expertise is crucial, as biological sciences are in continuous progress, requiring constant and continued education.

The use of test-enhanced learning with causal connection and in preparation for future learning has been used in health educational setting with positive results. However, most studies were performed in a controlled lab scenario and not in the "real world" of medicine classes, decreasing the external applicability of such experiments. Therefore, the aim of this study is to evaluate if a session of test-enhanced learning at the beginning of endocrinology course, using basic-clinical sciences connections of key concepts, would prepare for future learning of endocrinology on a theory-practical 4-week endocrinology course.

Methods Study design, participants and description of undergraduate endocrinology course This is a prospective, single center, non-blinded, RCT. Participants are students of medicine from Universidade Federal do Rio Grande do Sul (UFRGS), Brazil, in their third year of Medical School, recruited at the beginning of endocrinology undergraduate clinical placement. This clinical trial follows the Consolidated Standards of Reporting Trials (CONSORT) statement, which includes the completing the CONSORT checklist.

Sample size Based in a previous study, to find a difference in the percentage of correct answers in a cognitive test to evaluate retention of 12%, considering a SD of 26%, alpha error of 5%, beta error of 20%, and repeated assessments (baseline, 3 weeks and 6 months), 35 students will be necessary in each group. To account for possible losses of follow-up, 84 students will be included.

Study intervention All students will receive, in advance, a text with basic sciences information relevant to the learning of Endocrinology (supplementary material), with instructions to study the text before intervention day.

Students will be randomized to one of the interventions: TEL with questions about diabetes and adrenal (Block A, 6 questions) or thyroid and hypophysis (Block B, 6 questions). Important endocrinology concepts, such as fuel metabolism and circadian rhythm will be included in Block A, and feedback loops and hormone synthesis in Block B. Specific hormone functions will be part of both TEL Blocks.

Assessments At the same day of intervention, students will answer all questions 12 of the TEL session (questions from blocks A and B) with best answer multiple choice questions (immediate retention test). After 3 weeks and 6 months, the transfer of knowledge will be assessed with a 24 multiple choice questions test, based in clinical cases.

ELIGIBILITY:
Inclusion Criteria:

* Students will be consecutively invited to participated in the study before starting their Endocrinology placement and will be included after agreeing to participate and signing an informed consent

Exclusion Criteria:

* Students absent on the day of study intervention or on the four-week assessment will be excluded from analysis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
24 multiple choice questions test at 3 weeks | 3 weeks
  Scores in 24 multiple choice questions test to assess learning transfer from basic sciences to Endocrinology, in 3 weeks. This is an special designed test. It is not a scale. The score will be zero to 24. The highest score indicates the best performance.

SECONDARY OUTCOMES:
Immediate retention test | immediately after test
  Scores in immediate retention test (12 questions, in the same day as the TEL session)
24 multiple choice questions test at 6 months | 6 months
  Scores in 24 multiple choice questions test at 6 months
Metacognition questionnaires - professors | 4 weeks
  Results of metacognition questionnaires (not a scale)
Metacognition questionnaires - students | 4 weeks
  Results of metacognition questionnaires (not a scale)

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane B Leitao, MD, Principal Investigator — Hospital de Clínicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: No